CLINICAL TRIAL: NCT06442202
Title: Balanced Nutritional Diet Intervention on Body Composition Among Different FTO RS9939609 Gene in Obese Young Women In Bandung, Indonesia: A Randomised Controlled Trial
Brief Title: Balanced Nutritional Diet Intervention Among Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPB-202405.01
Record Dates: First submitted 2024-05-16; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obese Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Allele A + Diet Intervention (Experimental): Subjects with allele A carriers (AA/AT) FTO rs9939609 gene type, took a Balanced Nutritional Diet Intervention for 28 days. Besides, this group received nutritional education. Twelve (12) subjects were included in this group.
  Interventions: Dietary Supplement: Balanced Nutritional Diet; Behavioral: Nutritional Education
- T Homozygote + Diet Intervention (Experimental): Subjects with T homozygote FTO rs9939609 gene type, took a Balanced Nutritional Diet Intervention for 28 days. Besides, this group received nutritional education. Eight (8) subjects were included in this group.
  Interventions: Dietary Supplement: Balanced Nutritional Diet; Behavioral: Nutritional Education
- Allele A Control (Placebo Comparator): Subjects with allele A carriers (AA/AT) FTO rs9939609 gene type, control group, eat ad libitum. This group also received nutritional education. Ten (10) subjects were included in this group.
  Interventions: Behavioral: Nutritional Education
- T Homozygote Control (Placebo Comparator): Subjects with T Homogyzot FTO rs9939609 gene type, control group, eat ad libitum. This group also received nutritional education. Eight (8) subjects were included in this group.
  Interventions: Behavioral: Nutritional Education

INTERVENTIONS:
Dietary Supplement: Balanced Nutritional Diet — Food was provided during the intervention period 3 (three) times each day, i.e. breakfast, lunch and dinner. The food menu used a 30-day menu cycle. The characteristics of the Balanced Nutrition Diet that have been provided based on the distribution of the composition of the macronutrients that will be intervened in are as follows: 45-55% carbohydrates, 15-20% protein, and 20-25% fat (Ministry of Health 2014). The type of diet and portions that were given were the same for each menu unless there were certain food restrictions or allergies, and then the type of food was adjusted specifically to that individual. The calories that will be given range from 300-400 Cal for breakfast, 400-500 Cal for lunch, and 300-500 Cal for dinner.
  The choice of carbohydrates should be varied and prioritise complex carbohydrates such as whole grains. The choice of protein type is prioritised from low-fat protein sources and half of it is vegetable protein.
  Arms: Allele A + Diet Intervention; T Homozygote + Diet Intervention
Behavioral: Nutritional Education — Nutritional education is provided via online Zoom meetings with the help of educational media in the form of PowerPoint presentations/videos before entering the intervention period. The educational material that will be provided is regarding Guidelines for Balanced Nutrition, Food Safety, and Healthy Lifestyles (stress management and sleep time). The subject's understanding of the material provided was evaluated using an online quiz platform.

SUMMARY:
Food intake along with the gene are important factors that influence human nutrition status and health. Indonesia has a balanced nutrition diet guide for ideal food consumption. The FTO rs9939609 gene is known to be related to obesity. This study aimed to examine the effect of a balanced nutritional diet intervention on body composition among different single nucleotide polymorphisms (SNP) of the FTO rs9939609 gene in obese young women in Bandung City, West Java, Indonesia.

DETAILED DESCRIPTION:
A Balanced Nutrition Diet is a group of food menus that contain carbohydrates, fats, proteins, vitamins and minerals which are prepared based on the principles of diversity, balanced, regular and safe proportions in types and quantities that suit the body's needs adapted from the My Meal Dish Content/"Isi Piringku"; and "Tumpeng Gizi Seimbang" rule based on the Balanced Nutrition Guidelines of the Republic of Indonesia Minister of Health Regulation No. 41 year 2014. Although a balanced nutritional diet has not been widely used as a dietary intervention for obese people compared to the Mediterranean diet, there is research that shows that providing a low-calorie balanced nutritional diet based on traditional Indonesian food for 8 weeks can reduce body weight and body mass index, waist circumference, and body fat percentage of the research subjects were statistically significant.

Apart from eating habits, genetic factors also play an important role in the development of obesity. One of the most important genes associated with obesity is the FTO (fat mass and obesity-related) gene located on chromosome 16. Several polymorphisms in the FTO gene are known to be associated with increased body mass index (BMI) and other anthropometric values, severe obesity conditions, and risk of diabetes mellitus, although there are differences in different ethnicities. Several studies have also examined the association of the FTO gene with several parameters related to cardiovascular risk. The FTO rs9939609 gene polymorphism is one of the genes commonly studied in relation to obesity. The rs9939609 FTO gene consists of TT, TA, and AA genotypes. Allele A is a group of mutant genotypes or is called a risk allele (TA and AA) while TT is a group of wild genotypes or is considered a non-risk allele.

Evidence suggests that compared with TT wild type, the risk allele A FTO rs9939609 gene showed significantly higher body weight, body mass index, waist circumference, hip circumference, and waist-to-hip ratio. The waist-hip circumference ratio is a stronger indicator of cardiovascular disease than body mass index. The A allele carriers of the FTO rs9939609 polymorphism had a higher fat percentage. Until now, no one has ever linked the FTO gene polymorphism and the Balanced Nutrition Diet intervention, which is a reference in Indonesia, as well as its effect on the body composition of obese young women, especially in Sundanese ethnicity. This study aimed to examine the effect of a balanced nutritional diet intervention on body composition among 2 types of the FTO rs9939609 gene in obese young women in Bandung City, Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Obese women (fat percentage>35%) who had light to moderate physical activity based on PAL or who rarely exercised
* Sundanese ethnicity
* Aged 18-25 years
* Normal fasting blood glucose levels
* Willing to participate and sign an informed consent

Exclusion Criteria:

* Being pregnant and breastfeeding
* Had a history of chronic disease
* Regularly consuming antioxidant supplements and/or phytopharmaceuticals
* Currently participating in other research

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change of Body Compostition | 28 days
  Body composition will be measured twice, i.e. before randomization and 28 days after randomization. The measurement include body weight (kg); body height (cm); Body Mass Index (kg/m2); Waist circumference (cm); Hip circumference (cm); Waist-hip ratio; Visceral fat; Fat percentage (%); Resting metabolism (Cal); Total subcutaneous fat (%); Subcutaneous trunk (%); Subcutaneous arms (%); Subcutaneous legs (%); Total skeletal muscle (%); Skeletal trunk (%); Skeletal arms (%); Skeletal legs (%)

CONTACTS AND LOCATIONS:
Overall Officials: Prodi Gizi, Principal Investigator — Institut Pertanian Bogor
Locations (1):
- Prodi Gizi IPB, Bogor, Indonesia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT06442202/Prot_SAP_ICF_000.pdf